CLINICAL TRIAL: NCT05752955
Title: A Cluster-randomised Trial of a Complex Intervention to Reduce Anaemia and Cardiometabolic Risk During Pregnancy and in the First Year Following Birth in Women Living in Rural India (SMART Health Pregnancy 2)
Brief Title: SMART Health Pregnancy 2 - Intervention to Reduce Anaemia and Cardiometabolic Risk During Pregnancy and in the First Year Following Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 27-21
Record Dates: First submitted 2022-12-21; First posted 2023-03-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anemia of Pregnancy; Gestational Diabetes; Gestational Hypertension; Pre-Eclampsia; Anemia; Type 2 Diabetes; Hypertension
Keywords: Community Health Workers; mobile Health; Accredited Social Health Activist; Health Systems; Cardiometabolic diseases; Screening
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pre-Eclampsia; Anemia; Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor) The investigator and outcomes assessor will be blinded to allocation group. Each cluster will be coded and using a random number generator. The sites will only be unlinked after final database lock after endpoint adjudication for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMARThealth Pregnancy (Experimental): SMART Health Pregnancy is a complex intervention designed to be delivered on top of usual care. It comprises three parts:
  (i) A regular screening program focused on women's health during pregnancy and in the year following birth.
  (ii) An electronic decision support system (EDSS) (iii) An short messaging service (SMS) appointment reminder system
  Interventions: Other: SMARThealth Pregnancy
- Active Comparator: Usual Care (No Intervention): Usual antenatal and postnatal care. Women and health workers in the usual care clusters will not receive any additional support beyond that already offered under the local government programs

INTERVENTIONS:
Other: SMARThealth Pregnancy — At each visit, the CHW will:
  * Update history and contact details
  * Check haemoglobin with a point of care device.
  * Check BP
  * Check iron folic acid (IFA) supply and compliance
  * Brief screen for mental health problems
  An electronic decision support platform will provide advice if referral is needed. At the Primary Health Centre, doctor/s will be issued a tablet computer with a version of the SMARThealth Pregnancy App to:
  * Generate an automated list of all patients in the community who require review, with the dates of testing and referral, and with two-way communication back to the CHW.
  * Suggest management based on current Indian guidelines for the diagnosis and management of anaemia, hypertension and diabetes in pregnant and non-pregnant adults.
  Arms: SMARThealth Pregnancy

SUMMARY:
The goal of this clinical trial is to determine if a complex intervention called SMARThealth Pregnancy can improve the detection and management of high-risk conditions during pregnancy and in the first year after birth in women living in rural India.

The main questions it aims to answer are:

* Can screening of pregnant and postpartum women using the SMARThealth Pregnancy intervention decrease anaemia prevalence at 1 year after birth?
* Can the SMARThealth Pregnancy intervention improve postnatal testing after a pregnancy affected by hypertension and diabetes? Participants in the intervention group will be screened by their community health worker at several timepoints during pregnancy, and in the first year after birth using the SMARThealth Pregnancy tablet App. The community health worker will ask about each woman about her medical and obstetric history, then measure her blood pressure, haemoglobin (using a point of care device), and offer a referral for a glucose tolerance test when indicated. Women who screen positive for anaemia, hypertension or diabetes will be given advice and referred to the primary care doctor. The primary care doctor will have a complimentary tablet app to facilitate electronic referral and evidence-based prescribing when indicated. The comparison group will have usual antenatal and postnatal care.

DETAILED DESCRIPTION:
The primary aim of this study is to determine if the SMARThealth Pregnancy intervention can improve women's health in the year after pregnancy, specifically decrease the prevalence of anaemia by 9% and improve follow-up after a pregnancy affected by diabetes or hypertension. High glucose and blood pressure are the two leading contributors to cardiometabolic risk in women in India, thus it is hypothesised that targeting women identified in pregnancy at high risk of these conditions future risk can be decreased.

This study hypothesize SMARThealth Pregnancy intervention will:

* Decrease anaemia prevalence by 9% in women at 12 months after delivery by improving adherence to the current national government guidelines for iron folic acid supplementation through behavioural change interventions delivered to the woman by the Community Health Worker (CHW): (i) during pregnancy, with referral for iron sucrose injections where indicated; and, (ii) during breastfeeding, and (iii) after breastfeeding.
* Ensure women who develop gestational diabetes mellitus (GDM) are identified during pregnancy with appropriate referral, and followed up after birth and screened for the development of type 2 diabetes.
* Detect women with raised blood pressure during pregnancy, and provide ongoing periodic blood pressure (BP) monitoring after birth to detect ongoing hypertension.
* Provide all women during pregnancy and after birth regular mental health assessment and support leading to improved mental state and wellbeing
* Ensure after birth women are offered and have access to appropriate contraception choices
* Improve communication between different levels of the health system (community, subcenter, Primary health Centre (PHC) and district hospital)

Recruitment commenced in Siddipet district 6 June 2022 and will commence in Haryana 1 January 2023.

ELIGIBILITY:
Inclusion Criteria:

* For Primary health Centres:

  * located in the selected districts
  * provide pregnancy care
  * chief doctor (or equivalent) agrees to participate
* For women >12 weeks pregnant

Exclusion Criteria:

* women who plan to move away and not return to the same village for the next 12 months
* women unable to understand the local study language
* Women who do not give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3446 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change anaemia prevalence in women | 10-12 months after delivery
  Proportion of participants with any degree of anaemia (non-pregnant definition Hb < 12g/dL) between the intervention and control clusters

SECONDARY OUTCOMES:
Change the proportion of women with moderate and severe anaemia | 10-12 months after delivery
  Proportion of participants with moderate anaemia (Hb < 10g /dL) and severe anaemia (Hb < 8g /dL) between the intervention and control clusters
Postnatal screening for type 2 diabetes after GDM | 10-12 months after delivery
  Proportion of women with GDM who undergo screening for type 2 diabetes in the first year after delivery
Postnatal screening for hypertension after hypertensive disorder of pregnancy | 10-12 months after delivery
  Proportion of women with a hypertensive disorder of pregnancy screened for hypertension in the first year after delivery
Compliance with iron-folic acid supplements during pregnancy and breastfeeding | 10-12 months after delivery
  Self reported compliance with iron folic acid supplementation
De-worming treatment | during pregnancy
  Proportion of women during pregnancy who receive de-worming treatment
Point of care Haemoglobin (Hb) testing | 10-12 months after delivery
  Proportion of women who have a point of care Hb test during pregnancy and in the post natal period
Referral of high risk conditions | Six weeks post delivery
  The proportion of women detected with anaemia, hypertension or GDM correctly referred to primary or secondary care
Hypertension after hypertensive disorder of pregnancy | 10-12 months after delivery
  Differences in systolic and diastolic blood pressure in women who were diagnosed during pregnancy with hypertensive disorder of pregnancy
Dysglycaemia after a pregnancy affected by GDM | 10-12 months after delivery
  Difference in HbA1c, fasting and 2-hour glucose venous samples post 75 gram glucose load in those who developed GDM during pregnancy

OTHER OUTCOMES:
Differences in quality of life scores | 10-12 months after delivery
  Differences in EuroQuol 5D (EQ5D) score between baseline and at 12 months. The Five-item EQID uses scale of health score from 0 (worst imaginable) to 100 (best imaginable)
Differences in depression scores | 10-12 months after delivery
  Differences in Patient Health Questionnaire 9 (PHQ9) scores between baseline and at 12 months. Nine-item PHQ-9 use 4-point Likert-scaled items ranging from 0 (not at all) to 3 (nearly every day).
Differences in anxiety scores | 10-12 months after delivery
  Differences in Generalised Anxiety and Depression score 7 (GAD7) scores between baseline and at 12 months. The seven-item GAD-7 use 4-point Likert-scaled items ranging from 0 (not at all) to 3 (nearly every day).
Infant feeding | 6 weeks after delivery and 12 months after delivery]
  World Health Organization Infant and Young Feeding Assessment
Pregnancy intention | 10-12 months post natal
  Difference in London Measure of Unplanned pregnancy scores
Cost of care | 6 - 10 weeks after birth
  Direct and indirect costs of care during pregnancy and for the first six weeks after birth

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Hirst, MBBS MPH PhD, Principal Investigator — University of Oxford
Locations (1):
- The George Institute for Global Health, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual data and data dictionary will be made available for sharing on the day of publication of the main results.
  Data will be made available through a 3rd party data repository, via email request to the Principal Investigator on receipt of a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after publication of the main study findings and will be available for an indefinite period of time
Access Criteria: Data will be made available through a 3rd party data repository, via email request to the Principal Investigator on receipt of a signed data sharing agreement

REFERENCES:
- [Background] Nagraj S, Kennedy SH, Jha V, Norton R, Hinton L, Billot L, Rajan E, Arora V, Praveen D, Hirst JE. SMARThealth Pregnancy: Feasibility and Acceptability of a Complex Intervention for High-Risk Pregnant Women in Rural India: Protocol for a Pilot Cluster Randomised Controlled Trial. Front Glob Womens Health. 2021 May 28;2:620759. doi: 10.3389/fgwh.2021.620759. eCollection 2021. PMID 34816187
- [Derived] Hirst JE, Votruba N, Billot L, Arora V, Rajan E, Thout SR, Peiris D, Patel A, Norton R, Mullins E, Sharma A, Kennedy S, Jha V, Praveen D. A community-based intervention to improve screening, referral and follow-up of non-communicable diseases and anaemia amongst pregnant and postpartum women in rural India: study protocol for a cluster randomised trial. Trials. 2023 Aug 9;24(1):510. doi: 10.1186/s13063-023-07510-x. PMID 37559158
- See also: Study website — https://www.wrh.ox.ac.uk/research/smarthealth-pregnancy-improving-women2019s-life-long-health-in-rural-india